CLINICAL TRIAL: NCT02369380
Title: Volume Restoration of Plantar Pad With a Hyaluronic Acid Dermal Filler in Treatment of Metatarsalgia of Forefeet Further Use of High Heel Shoes
Brief Title: Volume Restoration of Plantar Pad With a Hyaluronic Acid Dermal Filler in Metatarsalgia
Acronym: ELFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.03.SPR.29108
Record Dates: First submitted 2014-12-09; First posted 2015-02-23 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2016-09

CONDITIONS: Metatarsalgia
MeSH Terms: conditions — Metatarsalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyaluronic acid (Experimental): Injections of hyaluronic acid under metatarsal heads
  Interventions: Device: Hyaluronic acid

INTERVENTIONS:
Device: Hyaluronic acid — Injections of Hyaluronic acid under the metatarsal heads

SUMMARY:
Aim of this study is to evaluate the decrease of plantar pain of forefeet due to restoration of plantar pad tissue density and of cushioning function with an hyaluronic acid dermal filler as mechanical-supplementation in subjects with metatarsalgia further use of high heel shoes

DETAILED DESCRIPTION:
This will be an open and single center study. There will be 4 study visits in total for each subject. Each subject will participate for a period of maximum 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female subject aged 30 years or older,
* Subject with pain sensation under metatarsal heads, further to use of high heels shoes at any moment of the day whatever the onset time,
* Subject with no previous injections under the metatarsal heads of forefeet.

Exclusion Criteria:

* Subject with a personal history of allergic/anaphylactic reactions including hypersensitivity to crossed-linked hyaluronic acid and to Lidocaine or amide local anesthetics
* Subject with cutaneous infection on either foot or with history of autoimmune diseases or auto-inflammatory diseases,
* Subject who wishes to wear orthotic supports (shock-absorbing insoles or arch supports, etc…).
* Subject with history of bleeding disorders or or erysipelas of the lower limbs,
* Subject with chronic inflammatory pain of the feet due to other non-mechanical causes, such as plantar fasciitis, arthritis, gout, Morton's neuroma.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pain assessment (Time to onset of pain (TInitial) (in hours) | Subject questioning at baseline after injections and change from baseline 1 month after baseline
  Time to onset of pain (TInitial) (in hours): duration between beginning of wearing high heel shoes and first pain sensations
Pain assessment (Time to maximum pain tolerance (TEnd) | Subject questioning at baseline after injections and change from baseline 1 month after baseline
  (in hours): duration between first pain sensations and the maximal pain tolerance (removing shoes).

SECONDARY OUTCOMES:
Podiatric criteria | Change from baseline 6 months after baseline
  Baro Podometric static examinations assessed by podiatrist at Baseline, 1 month, 3 months and 6 months after baseline to measure:
  - Mean pressure under metatarsal heads
Podiatric criteria (Baro Podometric static examinations) | Change from baseline 6 months after baseline
  Baro Podometric static examinations assessed by podiatrist at Baseline, 1 month, 3 months and 6 months after baseline to measure:
  - Maximum mean pressure under metatarsal heads

OTHER OUTCOMES:
Subject overall satisfaction | 6 months after baseline injections
  Overall satisfaction of subjects with injections outcome
Adverse Events | At each follow up visit:1 month, 3 months and 6 months after baseline
  Occurence of adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul Foumenteze, Dr, Principal Investigator
Locations (1):
- Dr Foumenteze, Cannes, France